CLINICAL TRIAL: NCT07338864
Title: A Post-market, Prospective, Observational Study to Evaluate Clinical Benefit, Performance and Safety of Cochlear™ Implants in an Adult Population: a Master Umbrella Investigation
Brief Title: A Study to Evaluate Clinical Benefit, Performance and Safety of Cochlear Implants in Adults
Acronym: ORBIT-MU
Status: Not yet recruiting | Type: Observational
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Other Study IDs: CLTD5819
Record Dates: First submitted 2026-01-04; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Hearing Loss; Hearing Implants
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Cochlear implant (CI1032): Participants implanted with a CI1032
  Interventions: Device: Cochlear Nucleus Nexa Cochlear implant (CI1032)
- Cochlear implant (CI1022): Participants implanted with a CI1022
  Interventions: Device: Cochlear Nucleus Nexa Cochlear implant (CI1022)
- Cochlear implant (CI1012): Participants implanted with a CI1012
  Interventions: Device: Cochlear Nucleus Nexa Cochlear implant (CI1012)

INTERVENTIONS:
Device: Cochlear Nucleus Nexa Cochlear implant (CI1032) — Participants will be implanted with a CI1032 cochlear implant as determined by the treating clinician
  Groups: Cochlear implant (CI1032)
Device: Cochlear Nucleus Nexa Cochlear implant (CI1022) — Participants will be implanted with a CI1022 cochlear implant as determined by the treating clinician
  Groups: Cochlear implant (CI1022)
Device: Cochlear Nucleus Nexa Cochlear implant (CI1012) — Participants will be implanted with a CI1012 cochlear implant as determined by the treating clinician
  Groups: Cochlear implant (CI1012)

SUMMARY:
The aim of this clinical investigation is to demonstrate the performance, clinical benefit and safety of commercial cochlear implant systems. Speech performance and subjective hearing results, and comparison with cochlear implant results available in literature, is intended to demonstrate the performance and clinical benefit of the cochlear implant systems investigated in this study.

ELIGIBILITY:
Inclusion criteria:

* Aged 18 years or older (at time of consent).
* Clinically established post-linguistic moderately severe to profound sensorineural hearing loss, in the ear to be implanted.
* Compromised functional hearing with hearing aid(s) or unlikely to receive benefit with hearing aid(s) in the ear to be implanted.
* Cochlear implant candidate as determined by the Principal Investigator. Meets local candidacy criteria for cochlear implantation.
* Candidate is a fluent speaker in the language used to assess speech perception performance.
* Willing and able to comply with study follow-up schedule.
* Willing and able to provide written informed consent.
* Candidate has access to a Smartphone compatible with Nucleus Smart App.

Exclusion criteria:

* Prior cochlear implantation in the ear to be implanted.
* Unrealistic expectations regarding the possible benefit, risks and limitations that are inherent to the surgical procedure and prosthetic device as determined by the investigator.
* Any contraindications for cochlear implantation listed in the relevant product physician's guide (to be specified per sub-investigation).
* Unable or unwilling to comply with the requirements of the clinical investigation as determined by the Investigator.
* Investigator site personnel directly affiliated with this study and/or their immediate families; immediate family is defined as spouse, parent, child or sibling.
* Cochlear employees or employees of Contract Research Organisations or contractors engaged by Cochlear for the purposes of this investigation.
* Women who are pregnant.
* Current participation, or participation in an interventional clinical study/trial in the past 30 days, involving an investigational drug or device (unless Cochlear sponsored and determined by Investigator or Sponsor to not impact this investigation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post lingually deafened adult adults who are a candidate for cochlear implantation.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Mean within-participant change in the word recognition score in quiet | Preimplantation to 6 months post-activation
  Percent correct word score from preimplantation to post-activation in the implanted ear.
  Score range: 0 to 100% correct, where a higher score is a better outcome.

SECONDARY OUTCOMES:
Incidence of adverse events and device deficiencies | From enrolment to 12 months post-activation
  Proportion of participants who experience an adverse event and the proportion of participants who experience a device deficiency
Mean within-participant change in Speech Spatial Qualities questionnaire (SSQ-12) | Preimplantation to 3, 6 and 12 months post-activation
  Speech, Spatial and Qualities of Hearing Scale Global Score (SSQ-12). Scores range from 0 to 10, where high scores indicate greater ability (less hearing disability).
Mean within-participant change in word recognition score in quiet | Preimplantation to 3 and 12 months post-activation.
  Percent correct word score from preimplantation to post-activation in the implanted ear. Score range: 0 to 100% correct, where a higher score is a better outcome.
Mean within-participant change in Living with Cochlear implants questionnaire (LivCI) | Preimplantation to 3, 6 and 12 months post-activation
  Living with Cochlear Implants Questionnaire (LivCI) evaluates the impact of a hearing device on four domains, Participation (range 0 to 12), Psychosocial & Wellbeing (range 0 to21), Stigma (range 0 to 15) and Management & Aesthetics (range 0 to 18), where a higher domain score indicates a positive patient report.
Mean within-subject change in speech recognition threshold in noise | 3, 6 and 12 months post-activation
  Speech reception threshold for a digit triplet test where 50% of the digits are correctly identified. The score upper limit is 20 dB, with no lower limit. A lower score indicates better performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Düsseldorf, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No